CLINICAL TRIAL: NCT06950918
Title: The Role of Flipped Classroom and Flip-Jigsaw in Theoretical Physiotherapy Education: A Comparison of Knowledge, Motivation and Engagement
Brief Title: Flipped Classroom vs. Flip-Jigsaw in Theoretical Physiotherapy Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Collaborators: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ziya Yildiz, Dr. PhD (physiotherapy and rehabilitation), Isparta University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: postdr2
Record Dates: First submitted 2025-03-21; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Physiotherapy and Rehabilitation; Educational Technology; Educational Interventions; Students; Undergraduate Health Professional Students
Keywords: Flipped Clasroom; Flip-J; Learning Model; Physiotherapy education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flipped Clasroom Group (Experimental): Pre-class: Asynchronous video lectures covering theoretical content (e.g., public health principles, manual therapy techniques) were provided via an online platform. Students were required to review materials before in-person sessions. In-class: Instructor-led interactive discussions, case analyses, and problem-solving activities focused on applying theoretical knowledge. No peer-teaching components were included. Structure: Emphasis on self-paced learning followed by collaborative, instructor-guided reinforcement.
  Interventions: Other: Experimental
- Flipped-Jigsaw Group (Experimental): Pre-class: The same video lessons as the FC group are delivered only to the students in the expert group in the pre-class content delivery.
  In-class: Structured peer-teaching using the Jigsaw technique:
  Expert Groups: Students were divided into small groups, each assigned a subtopic (e.g., cervical spine assessment techniques) to master.
  Home Groups: Students returned to mixed groups to teach their subtopic to peers, ensuring collective knowledge integration.
  Instructor Role: Facilitated discussions and provided feedback but did not lead content delivery.
  Structure: Combines self-paced learning with peer-driven, collaborative skill-building.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — This study is a quasi-experimental parallel group design comparing Flipped Classroom (FC) and Flip-Jigsaw models in a theoretically-oriented public health course. Both groups used the same pre-prepared video lectures to standardize content, but differentiated in-class strategies: The FC group used instructor-led discussions, while the Flip-Jigsaw group used Jigsaw technique and peer teaching (students learning subtopics in "expert groups" and teaching them in "master groups"). Unlike traditional FC, this hybrid model includes systematic peer collaboration and role-based accountability mechanisms. Theoretical knowledge acquisition, motivation and engagement outcomes were assessed through quantitative tests (pre-post-retention tests) and qualitative interviews, and objectivity was ensured in practical exams with single-blinded assessors. The study brings innovation to the literature as it is the first study to demonstrate the unique effect of Flip-Jigsaw in theoretical courses in the fie

SUMMARY:
Study Summary:

This quasi-experimental pre-test-post-test study aims to compare the effects of Flipped Classroom (FC) and Flip-Jigsaw instructional models on theoretical knowledge acquisition, academic motivation, and class engagement among 86 third-year physiotherapy undergraduates enrolled in a theory-based public health course.

Primary Questions:

How does the hybrid Flip-Jigsaw model impact learning and motivation outcomes compared to FC alone?

Do FC and Flip-Jigsaw differ in enhancing theoretical knowledge, motivation, and participation?

Comparison: Researchers will compare the FC group (pre-class videos + in-class discussions) with the Flip-Jigsaw group (video-based pre-learning + structured peer teaching) to evaluate differences in outcomes.

Participant Tasks:

Attend lectures and complete pre-/post-knowledge tests.

Engage in practical sessions (FC: group discussions; Flip-Jigsaw: peer-led jigsaw activities).

Complete motivation surveys and participation assessments.

Significance: Addresses the gap in understanding Flip-Jigsaw's efficacy in physiotherapy education, despite prior reports on FC and Jigsaw's individual benefits.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-25
* Volunteering to participate in the study
* Taking the course for the first time
* Having access to the Internet
* Compulsory course attendance

Exclusion Criteria:

* Being a minor student
* Not being the first undergraduate education
* To have previously attended courses, seminars, webinars, etc. related to public health
* Participation in other pedagogical studies during the same academic term.
* Failure to complete ≥1 assessment (pre-test, post-test, or surveys).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Level of theoretical knowledge | pre-test and immediately after the intervention (7 weeks after study enrollment)
  The theoretical knowledge part of the course content will be done with a 20-question 5-choice multiple choice test. The same multiple choice test will be used as a post test after the lecture.
Level of motivation | immediately after the intervention (7 weeks after study enrollment)
  The adapted Instructional Material Motivation Scale was administrated to measure the participants' motivation towards the instructional material . The scale consists of 36 five-point Likert scale items covering four sub-scales.
Level of student engagement | immediately after the intervention (7 weeks after study enrollment)
  Course duration can be recorded in minutes on the education platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Raw data and statistical analyses can be shared, with participant identities obscured.
Supporting Information: SAP